CLINICAL TRIAL: NCT05459025
Title: Effectiveness of Aromatherapy Yoga in Stress Reduction and Sleep Quality Improvement Among Female College Students: A Quasi-Experimental Study
Brief Title: Effectiveness of Aromatherapy Yoga
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yang Shang-Yu (Other)
Responsible Party: Sponsor-Investigator, Yang Shang-Yu, Assistant professor, National Cheng Kung University
Organization: National Cheng Kung University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HZAUHU-2021-0001
Record Dates: First submitted 2022-07-12; First posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Female College Students
MeSH Terms: interventions — Yoga

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aromatherapy yoga (Experimental): Each intervention session lasted 90 min, between 6 p.m. and 7:30 p.m. The course was held in a yoga classroom once a week, in an area of 30 m × 35 m. Furthermore, the total intervention period lasted for 12 weeks.
  Interventions: Behavioral: Aromatherapy yoga
- Yoga (Active Comparator): Each intervention session lasted 90 min, between 6 p.m. and 7:30 p.m. The course was held in a yoga classroom once a week, in an area of 30 m × 35 m. Furthermore, the total intervention period lasted for 12 weeks.
  Interventions: Behavioral: Yoga

INTERVENTIONS:
Behavioral: Aromatherapy yoga — The research assistant diluted the Lavandula angustifolia essential oil with distilled water (1:75) 10 min before the yoga session started. The solution was then atomized by three aroma diffusers, placed in the front, middle, and back of the classroom. The distance from each participant was less than 10 m to ensure that the aroma was absorbed com-pletely. The yoga course for the aromatherapy yoga group was the same as that of the yoga only group. The yoga group only took a yoga course, without aromatherapy.
  Arms: Aromatherapy yoga
Behavioral: Yoga — The design of the yoga lessons was based on a past study and a professional yoga instruction book. Yoga lessons were led by certified yoga tutors.
  Arms: Yoga

SUMMARY:
College students, particularly female students, often suffer from severe stress and poor sleep. Aromatherapy yoga has become a popular exercise in recent years and may help reduce stress and improve sleep quality, although empirical evidence is limited. We investigated the effective-ness of aromatherapy yoga intervention in reducing stress and improving sleep quality among female college students. Eighty-nine participants (44 in the experimental group [aromatherapy yoga] and 45 in the control group [yoga]), with an average age of 19.88 ± 1.13 years, were en-rolled in this quasi-experimental study. Interventions were performed in the respective groups once a week for 12 weeks, for 90 minutes each time. The Wilcoxon signed-rank test and Mann-Whitney U test (including effect size) were used to test the differences in stress reduction and sleep quality before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* We included female college students aged > 18 years, who were able to understand the questionnaire.

Exclusion Criteria:

* We excluded male students, those with a history of respiratory disease, asthma, or allergy to flowers, plants, or essential oils, those who worked at night, and those with a history of mental diseases.

Ages: 18 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 89 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale 14 (PSS-14) | 10-15 minutes
  PSS-14 is the scale that is most widely used for measuring the degree to which situations in one's life are appraised as being stressful.
Pittsburgh Sleep Quality Index (PSQI) | 10-15 minutes
  The PSQI developed by Buysse et al. [45], which evaluates sleep quality of the participants in the past month.

CONTACTS AND LOCATIONS:
Locations (1):
- Asia Univeraity, Taichung, WuFeng, Taiwan